CLINICAL TRIAL: NCT03978728
Title: Analysis of Endotoxin Activity in Patients With Extracorporeal Membrane Oxygenation Life Support System
Brief Title: Analysis of Endotoxin Activity in Patients With ECMO
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201811061RINC
Record Dates: First submitted 2019-06-02; First posted 2019-06-07 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Shock; Respiratory Failure
MeSH Terms: conditions — Shock, Cardiogenic; Respiratory Insufficiency | interventions — Ex utero Intrapartum Treatment Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO patients: Patients with ECMO support
  Interventions: Device: Extra-corporeal membrane oxygenation

INTERVENTIONS:
Device: Extra-corporeal membrane oxygenation — Cardiovascular shock patients received extra-corporeal membrane oxygenation suppot.

SUMMARY:
Extra-corporeal membrane oxygenation (ECMO) can temporarily help patients gain time to wait for cardiopulmonary recovery or further treatment in patients with cardiopulmonary failure. Whether the blood flow provided by the ECMO can maintain the perfusion of various organs is an important factor affecting survival. Some ECMO patients died after the complication of sepsis. Our previous pilot analysis has recognized several ECMO patients with complicated sepsis has high endotoxin activity level. Endotoxemia can also occur in heart surgery and after cardiopulmonary bypass, trauma, organ transplantation, and out-of-hospital cardiac arrest patients. These trials used endotoxin activity analysis (EAA, EAATM, Spectral Diagnostics Inc., Canada) to analyze endotoxin activity. In addition, studies have indicated that the combination of procalcitonin (PCT) concentration and EAA activity can improve the accuracy of predicting sepsis. The primary aim of this study is to detect endotoxin activity in patients with ECMO support and compare whether the prognosis was associated with different level of EAA activity. The secondary aims are to analyze the risk factors leading to high EAA activity and investigate the diagnostic value of septic shock combining PCT examination. We suggest that the results of this study may help the ECMO medical team identify patients at high risk for septic shock and conduct adequate managements to improve patient survival and quality of life after survival.

ELIGIBILITY:
Inclusion Criteria:

* patients with ECMO support

Exclusion Criteria:

* < 20 years old or > 90 years old
* not be able to collect blood sample within 48 hours after placement of ECMO
* change plan to palliative care and plan to remove ECMO
* non-native speakers

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitents with extra-corporeal membrane oxygenation support
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Endotoxin activity level | within 48 hours
  Endotoxin activity level is measured by endotoxin activity analysis kit

SECONDARY OUTCOMES:
Endotoxin activity level | within 24 hours
  Endotoxin activity level is measured by endotoxin activity analysis kit
Endotoxin activity level | within 72 hours
  Endotoxin activity level is measured by endotoxin activity analysis kit
Endotoxin activity level | within 96 hours
  Endotoxin activity level is measured by endotoxin activity analysis kit
Procalcitonin level | within 48 hours
  Procalcitonin level in ECMO patients
Cystatin C level | within 48 hours
  Cytatin C level in ECMO patients
Diamine oxidase level | within 48 hours
  Diamine oxidase level in ECMO patients

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No